CLINICAL TRIAL: NCT00891475
Title: Phase II Trial of Palliative Radiofrequency Ablation in Metastatic Renal Cell Carcinoma Patients With Small Primary Tumor
Brief Title: Palliative Radiofrequency Ablation in Metastatic Renal Cell Carcinoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kidney Cancer Research Bureau (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCRB-003
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Carcinoma, Renal Cell
Keywords: metastatic renal cell carcinoma; radiofrequency ablation
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Radiofrequency Ablation; Interferon-alpha; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): 38 patients
  Interventions: Procedure: Radiofrequency ablation; Interferon-alpha
- Arm 2 (Experimental): 38 patients
  Interventions: Procedure: Radiofrequency ablation; Sunitinib maleate
- Arm 3 (Experimental): 38 patients
  Interventions: Drug: Sunitinib maleate

INTERVENTIONS:
Procedure: Radiofrequency ablation; Interferon-alpha — Patients undergo ablation by radiofrequency energy under CT-guidance. RFA continues until the entire tumor is treated. Treatment ceases when the entire lesion has undergone necrosis or the zone of necrosis or significant heat deposition approaches vital neurovascular structures. 38 patients will receive following immunotherapy with Interferon-alpha 9 MIU subcutaneously three times per week, 3 weeks on, 3 weeks off till progression. 38 patients will receive sunitinib maleate 50 mg orally once day, 28 days on, 14 days off till progression. Evaluation for response will be after second cycle.
  Arms: Arm 1
Procedure: Radiofrequency ablation; Sunitinib maleate — Patients undergo ablation by radiofrequency energy under CT-guidance. RFA continues until the entire tumor is treated. Treatment ceases when the entire lesion has undergone necrosis or the zone of necrosis or significant heat deposition approaches vital neurovascular structures. 38 patients will receive sunitinib maleate 50 mg orally once day, 28 days on, 14 days off, till progression. Evaluation for response will be after second cycle.
  Arms: Arm 2
Drug: Sunitinib maleate — 38 patients with unresected primary tumor will receive sunitinib maleate 50 mg orally once day, 28 days on, 14 days off, till progression. Evaluation for response will be after second cycle.
  Arms: Arm 3

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of Radiofrequency ablation in metastatic renal cell carcinoma patients with primary tumor less than 5 cm before medical treatment. Ablation may allow for reduced morbidity and may increase the likelihood of patients receiving systemic therapy.

DETAILED DESCRIPTION:
Nephrectomy has become an integral part of the management of patients with metastatic kidney cancer. Performing nephrectomy in these patients is not without risk, however. The very real chance of significant metastatic disease progression during the postoperative period or complication before or during surgery that may prolong postoperative recovery could potentially delay or prevent the administration of systemic therapy in the postoperative period. Patient selection for surgery remains critical for success.

Radiofrequency ablation (RFA) is a medical procedure where tumor is ablated using microwave energy to treat a medical disorder. The benefits of RFA in selected metastatic renal cell carcinoma patients with small primary tumor (<5 cm) will be evaluated in this Phase I/II study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven renal cell carcinoma before RFA;
* Primary tumor no grater than 5 cm;
* CT-confirmed metastatic measurable sites;
* Good prognosis by adapted MSKCC criteria;
* No treatment for RCC;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2008-05; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 11 months

SECONDARY OUTCOMES:
Overall survival | 24 months
rate of complications | 1 year
time from the end of ablation to start of medical treatment | 3 months
Progression-free survival | 6 months
Quality of life (QOL) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ilya V. Tsimafeyeu, MD, Study Director — KCRB; Bin Chung, MD, Principal Investigator — Beijing Hospital
Locations (1):
- Ilya Tsimafeyeu, Moscow, Russia